CLINICAL TRIAL: NCT03120962
Title: Effect of Early Use of Oxycodone During the Acute Phase of Herpes Zoster on Preventing Postherpetic Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-012
Record Dates: First submitted 2017-04-16; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Herpes Zoster; Post-herpetic Neuralgia
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Oxycodone; Gabapentin; Famciclovir

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oxycodone (Experimental): Oxycodone 20mg/day, for 4 weeks and famciclovir 500mg three-times daily for 7 days.
  Interventions: Drug: Oxycodone; Drug: Gabapentin; Drug: Famciclovir
- standard treatment (Active Comparator): Gabapentin 900mg/day, titrated up to max tolerated dose or 1800mg/day (whichever is lower), for 4-12 weeks and famciclovir 500mg three-times daily for 7 days.
  Interventions: Drug: Gabapentin; Drug: Famciclovir

INTERVENTIONS:
Drug: Oxycodone — Oxycodone 20mg/day, for 4 weeks
  Other Names: Oxycontin
  Arms: oxycodone
Drug: Gabapentin — Gabapentin 900mg/day, titrated up to max tolerated dose or 1800mg/day, for 4-12 weeks
  Other Names: neurontin
Drug: Famciclovir — Famciclovir 500mg three-times daily for 7 days
  Other Names: Famvir

SUMMARY:
Postherpetic neuralgia (PHN) which persists more than 90 days after the resolution of the acute shingles episode is the most common complication of herpes zoster. The continued pain or paresthesia not only affects patient quality of life, but also causes physical disability, emotional distress and social isolation. Conventional treatments for PHN are only partially work in some patients or not work at all in others. Once PHN presences, it is often refractory to the treatment, therefore, it is important to prevent the occurrence of PHN. In the study, the investigators want to identift whether the additional use of oxycodone therapy to current standard treatment in acute herpes zoster patients will decrease the incidence of post-herpetic neuralgia.

DETAILED DESCRIPTION:
Herpes zoster (HZ) results from reactivation of the latent varicella zoster virus in sensory ganglia, with characteristic symptom of painful skin rash and localized blisters. Usually, the rash heals and pain resolves within two to four weeks, but in some patients the pain continues to persist for more than 90 days after the onset of rash, which is known as postherpetic neuralgia (PHN).

PHN is the most common complication of HZ. Depending on the definition, the incidence of HZ patients developing PHN varied from approximately 5% to 30%. The continued pain or paresthesia not only affects patient quality of life, but also causes physical disability, emotional distress and social isolation. Conventional treatments for PHN include topical lidocaine or capsaicin, anticonvulsants, tricyclic antidepressants, and opioids. However, whether prescribed alone or in combination, these medications are only partially work in some patients or not work at all in others. Once PHN presences, it is often refractory to the treatment, therefore, it is important to prevent the occurrence of PHN. Previous studies have identified age, rash duration before consultation, presence of severe rash and acute pain severity as predictors of increased PHN risk. Thus, the treatment of acute pain of herpes zoster has the potential to prevent the development of PHN.

Acute zoster pain represents a combination of nociceptive and neuropathic pain which can be relieved by oxycodone. However, it is not known whether the additional use of oxycodone therapy to current standard treatment in acute herpes zoster patients will decrease the incidence of post-herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

Provide written informed consent. Male or female patients of 50 years of age and older. Diagnosis of uncomplicated herpes zoster presenting within the first 7 days of vesicles.

Average pain score pre-therapy greater or equal than 4 on a 0-10 visual analogue scale (VAS; 0 = no pain; 10 = worst possible pain).

Exclusion Criteria:

Patients with a history of chronic pain. Patients with immune dysfunction including congenital immune deficiency, active malignancy of any type, collagen vascular diseases, organ or bone marrow transplantations, known infection with HIV or severe atopic dermatitis.

Patients who have received cytotoxic drugs or immunosuppressive therapy (e.g., chronic systemic corticosteroids) within the previous 3 months.

Patients who have received systemic anti-VZV medications or immunomodulatory medications (including interferon) within the previous 4 weeks.

Patients with impaired renal function: calculated creatinine clearance of <30 mL/min using Cockcroft and Gault formula.

Patients with abnormal liver function (alanine transaminase (ALT) or aspartate;transaminase (AST) levels greater than five times the upper limit of the normal range).

Patients with a history of intolerance or hypersensitivity to acyclovir, penciclovir, valacyclovir, famciclovir, gabapentin or oxycodone.

Patients with alcohol or drug abuse history within the previous 5 years. Patients currently receiving therapy with opioid analgesics or tramadol. Patients currently receiving therapy with gabapentin or tricyclic antidepressants.

Pregnant females and nursing mothers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with zoster pain. | 3 months
  proportion

SECONDARY OUTCOMES:
Proportion of patients with zoster pain | 6 months and 1 year
  proportion
Pain intensity | 3 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months and 6 months
  0-10 visual analogue scale (VAS; 0 = no pain; 10 = worst possible pain)
Quality of life | 3 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months and 6 months
  zoster brief pain inventory
Side-effects | 3 days, 7 days, 2 weeks, 3 weeks, 1 month, 3 months and 6 months
  proportion of side effects

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dworkin RH, Barbano RL, Tyring SK, Betts RF, McDermott MP, Pennella-Vaughan J, Bennett GJ, Berber E, Gnann JW, Irvine C, Kamp C, Kieburtz K, Max MB, Schmader KE. A randomized, placebo-controlled trial of oxycodone and of gabapentin for acute pain in herpes zoster. Pain. 2009 Apr;142(3):209-217. doi: 10.1016/j.pain.2008.12.022. Epub 2009 Feb 4. PMID 19195785